CLINICAL TRIAL: NCT00738634
Title: IN2SHAPE Intervention to Stay Healthy and Physical Everyday: A Randomised Controlled Trial for the Feasibility and Effectiveness of a Self-motivated Physical Activity Intervention on the Mental Health of Adolescents.
Brief Title: IN2SHAPE: A Study of Physical Activity and Depressive Symptoms in Adolescence
Acronym: IN2SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Australian National University (Other)
Responsible Party: Principal Investigator, Jacqui Brewer, Ms, Australian National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008/008 HREC
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Depression; Motor Activity; Adolescent
MeSH Terms: conditions — Depression; Motor Activity | interventions — Nutritional Status

ARMS (3):
- Physical activity mediated (Experimental): Self-motivated physical activity intervention
  Materials mailed to participants
  Interventions: Behavioral: Self-motivated physical activity
- Nutrition control (Active Comparator): Nutrition attention-control arm.
  Delivered by researcher.
  Interventions: Behavioral: Nutrition
- Physical activity researcher contact (Experimental): Self-motivated physical activity intervention
  Delivered by researcher.
  Interventions: Behavioral: Physical activity researcher contact

INTERVENTIONS:
Behavioral: Self-motivated physical activity — Components:
  1. Physical activity education in the form of a brief booklet (double sided A4 page).
  2. Physical activity motivation tips (one sided A4 page).
  3. Pedometer
  4. Monitoring chart
  5. Online presentation of common obstacles and ways to overcome these obstacles
  Arms: Physical activity mediated
Behavioral: Nutrition — Components:
  1. Nutrition education booklet (Double-sided A4 page)
  2. Nutrition motivation tips (single-sided A4 page)
  3. Nutrition monitoring chart
  4. Online presentation of common obstacles and ways to overcome these obstacles
  Arms: Nutrition control
Behavioral: Physical activity researcher contact — Behavioral: Self-motivated physical activity
  Components:
  1. Physical activity education in the form of a brief booklet (double sided A4 page).
  2. Physical activity motivation tips (one sided A4 page).
  3. Pedometer
  4. Monitoring chart
  5. Online presentation of common obstacles and ways to overcome these obstacles
  Arms: Physical activity researcher contact

SUMMARY:
The purpose of this study is to determine whether physical activity prevents development of depressive symptoms in adolescents.

DETAILED DESCRIPTION:
The primary objective of the project is to establish whether increasing physical activity can promote mental well-being in adolescents who are already displaying some depressive symptoms.

A further objective is to evaluate the feasibility of a novel self-motivated physical activity intervention, which has been designed for this project.

The final objective of this project is to investigate alternative intervention delivery modes, for an adolescent sample with subclinical depressive symptomatology, i.e., presenting with some depression symptoms but not at a level where major depressive disorder would be diagnosed. We aim to compare the effect of a completely mediated delivery approach for physical activity (i.e., no researcher contact) and a mediated intervention with face-to-face contact and fortnightly check-in telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents from Grades 7-10 (high school) and their parents/guardians.
* Adolescents scoring in the middle range (14-30) on the Centre for Epidemiological Studies-Depression Scale (possible range 0-60).

Exclusion Criteria:

* Adolescents currently engaging in 60+ minutes of physical activity per day.
* Adolescents who have experienced psychosis, schizophrenia or bipolar disorder.
* Adolescents who score >30 on the CES-D (indicator of severe depression).
* Adolescents who have physical health problems or conditions which preclude them from participation in regular physical activity.
* Lack of written consent from adolescent and/or parent guardian.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Depression as measured by the Centre for Epidemiological Studies-Depression Scale (CES-D) | Baseline, 8 weeks and 4 month post-intervention follow-up
Physical activity levels | Baseline, 8 weeks and 4 month post-intervention follow-up

SECONDARY OUTCOMES:
Anxiety (RCMAS) | Baseline, 8 weeks, and 4 month post-intervention follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline L Brewer, BPsyc Hons, Principal Investigator — The Australian National University; Janine Walker, PhD, Study Chair — The Australian National University; Prof Helen Christensen, PhD, Study Director — The Australian National University
Locations (1):
- The Centre for Mental Health Research, Canberra, Australian Capital Territory, Australia